CLINICAL TRIAL: NCT04944719
Title: Pneumococcal Nasopharyngeal Colonization as Predictor of Community-Acquired Pneumonia in Adults With Chronic Diseases: A Real-word Evidence, Prospective, Observational, Multicenter, Cohort Study.
Brief Title: Pneumococcal Nasopharyngeal Colonization as Predictor of Community-Acquired Pneumonia (CAP) in Adults With Chronic Diseases.
Acronym: CAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de la Sabana (Other)
Responsible Party: Sponsor
Other Study IDs: MED-285-2020
Record Dates: First submitted 2021-06-10; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Streptococcus Pneumoniae Pneumonia; Streptococcus Pneumoniae Infection; Streptococcus Pneumoniae Infection Invasive; Community-acquired Pneumonia
Keywords: Streptococcus pneumoniae (neumococo); Community Acquired Pneumonia (CAP); Nasopharyngeal colonization; Serotypes; Adults with Chronic Diseases
MeSH Terms: conditions — Pneumonia; Pneumococcal Infections; Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — blood, nasopharyngeal aspirate, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chronically ill adult patients colonized by streptococcus pneumoniae: At baseline, adult patients with chronic disease who are colonized with Streptococcus pneumoniae will be identified. Then, after determining the colonized subjects, monthly telephone follow-up and clinical outcome will be determined to identify patients who develop CAP or IPD. Additionally, follow-up samples similar to baseline will be taken to determine colonization by other serotypes or resolution of colonization status in these patients.
  Interventions: Diagnostic Test: nasopharyngeal aspirate
- chronically ill adult patients not colonized by streptococcus pneumoniae: Subjects who are not colonized with S. pneumoniae will be followed by monthly telephone follow-up and clinical outcome will be determined to identify patients who develop CAP or IPD. Additionally, follow-up samples similar to baseline will be collected every six months to determine colonization during the follow-up time in the study.
  Interventions: Diagnostic Test: nasopharyngeal aspirate

INTERVENTIONS:
Diagnostic Test: nasopharyngeal aspirate — nasopharyngeal aspirate to determinate colonization by streptococcus pneumoniae

SUMMARY:
Streptococcus pneumoniae (pneumococcus) is a commensal bacterium, often isolated in the nasopharynx of preschool children and older adults with weakened immune systems, a pathogen that remains the leading cause of Community-Acquired Pneumonia (CAP) and invasive pneumococcal disease (IPD) such as Sepsis and Meningitis.

CAP is the sixth leading cause of overall mortality and the first cause of infectious disease in Colombia and the world (Montúfar et al, 2013; GBD, 2016; WHO, 2018), and both its incidence and prevalence have remained stable over the past 3 decades. Likewise, CAP due to S. pnemoniae is the most common cause of lower respiratory tract infections in humans worldwide and is associated with high morbidity and mortality in patients who suffer from it.

Pneumococcus frequently colonizes the nasopharynx of children and adults and, therefore, this condition has been postulated as a risk factor for the development of CAP. There are reports of the effect of nasopharyngeal colonization in infants, but the implications of this colonization in adults, especially adults with chronic comorbidities, are not known.

Additionally, several studies point to a relationship between pathogenicity, colonization capacity, and disease severity according to the infecting pneumococcal serotype. Therefore, it is not known which pneumococcal serotypes are most frequently colonized by adults with chronic diseases (cardiovascular disease (CVD), chronic obstructive pulmonary disease (COPD), renal disease (RHD), rheumatological disease (MDR), Diabetes Mellitus (DM), among others) and the potential clinical implications of this colonization.

For these reasons, this research aims to study the phenomenon of colonization by pneumococcus in patients with chronic diseases for the development of CAP, and the relationship between the virulence genes of different serotypes and the outcome in invasive pneumococcal disease (IPD).

This study is based on real evidence (from clinical practice) and translational medicine, is prospective-observational, multicenter and cohort type in consecutive patients. Thus, in a first phase the clinical observation of the subjects will be carried out, a second phase of follow-up and sampling in the patients, and a third phase of molecular analysis.

DETAILED DESCRIPTION:
Streptococcus pneumoniae (the pneumococcus) is responsible for more than 5 million deaths a year globally (Aliberti et al., 2016; Reyes et al., 2017). This opportunistic Gram-positive bacterium is the most frequently identified bacteria in patients with CAP, acute meningitis, and otitis in children and adults (Paterson et al., 2010; Hinojosa et al., 2014).

The pneumococcal disease has changed during the last decade due to universal pneumococcal vaccination programs, especially in children, patients with chronic pulmonary diseases, and patients older than 65 years old. Now, serotypes thought to be not clinically significant are frequently identified in patients with pneumococcal diseases (Imohl et al., 2015; Vlachopoulos et al., 2015; Cilloniz et al., 2016; Diao et al., 2016; Suzuki et al., 2017).

However, mortality and morbidity associated with pneumococcal infection in adults have remained relatively steady during the last decades (Jain et al., 2015; Bellew et al., 2018; Wunderink et al., 2018). Several hypotheses have been generated to explain this phenomenon. Among the most studied, researchers have documentedthat circulating pneumococcal serotypes are different now, and thus, currently available vaccines may not be as useful to prevent invasive pneumococcal diseases now (Aliberti et al., 2013; Cilloniz et al., 2016).

Moreover, adults are not frequently vaccinated with the pneumococcal vaccine, and only a very restrictive group of patients receive the vaccine. In Colombia, it is not known whether even that restrictive group of adults with an indication for a pneumococcal vaccine have been vaccinated, following national and international guidelines. More importantly, it is unknown whether other groups of patients with chronic medical diseases might benefit from receiving this vaccine.

Importantly, it is also unknown, which are the most prevalent serotypes causing colonization and invasive infections in adults with chronic diseases in Colombia.

We have recently carried out a multicenter, multinational, worldwide study designed to characterize better the etiology of CAP (the most frequent infection caused by the pneumococcus) (Aliberti et al., 2016; Carugati et al., 2016; Gramegna et al., 2018; Restrepo et al., 2018; Radovanovic et al., 2019).

In this study, we enrolled more than 3,700 patients in six continents, finding that S. pneumoniae continues to be the most frequent bacterial pathogen identified in patients with CAP worldwide. However, in this study, we also documented that the pneumococcal vaccination rate is meager (data not yet published). Thus, we firmly believe that identifying whether pneumococcal vaccination is adequate in our country (Colombia), and more importantly, which are the most prevalent pneumococcal serotypes colonizing the nasopharyngeal epithelium of patients with chronic medical conditions, might help us to identify new indications for pneumococcal vaccination and to help decrease the burden of pneumococcal diseases.

Therefore, here we will attempt to provide new information to characterize better pneumococcal nasopharyngeal colonization of patients with chronic medical diseases, its implications, its overtime dynamics, and how this colonization might be associated with CPA development. Moreover, here we will be able to characterize vaccination compliance and how this previous vaccination might modify the natural course of pneumococcal disease (i.e., nasopharyngeal colonization precedes pneumococcal pneumonia). Finally, here we will carry out real-world evidence, prospective study evidence that will provide generalizable data for clinicians around the globe.

This is real-world evidence, prospective, observational, multicenter, a cohort study of consecutive patients.

Inclusion Criteria

All consecutive ambulatory patients that assist to 5 outpatient clinics with chronic diseases such as heart failure, HBP, chronic cardiac arrhythmias, rheumatic diseases, non-cystic-fibrosis bronchiectasis, COPD, among others, with the following inclusion criteria will be included in the study:

* Older than 18 years old
* Patients assisting to cardiology, pulmonology, endocrinology or rheumatology clinic in participating centers
* Patients in whom vaccination information is available and confirmed in the medical records (this information will also be confirmed during the patient's interview)
* Patients that sign informed consent form.

Exclusion Criteria

* Patients diagnosed with CAP during the past 90 days
* Patients admitted to the hospital during the last 7 days
* Patients with limitation to provide biological samples

Baseline procedures

After identifying potential study subjects, informed consent will be obtained for interested patients, and a unique identification number will be assigned for each study' participant. Under any circumstance, patients will receive more than one identification number. Then, demographic data, past medical history, comorbid conditions, recent hospitalization, and biological samples will be gathered.

We will perform a nasopharyngeal swap to identify which patients are colonized with S. pneumoniae and to identify which are the most prevalent pneumococcal serotypes. We will draw 20cc of blood to identify inflammatory biomarkers, and 30cc urine samples will be collected for laboratory analyses.

Biological samples processing

After collecting samples in ambulatory clinics during study visits, these will be referred to our centralized research laboratory localized in the Universidad de La Sabana to carry out laboratory experiments. All nasopharyngeal swaps will be culture for pneumococcal identification; if S. pneumoniae is identified, we will characterize in our laboratory pneumococcal serotypes. Moreover, we will perform rtPCR to better identify and quantify pneumococcal colonization in the nasopharyngeal swabs.

We will also quantify serum biomarkers of inflammation, using commercially available ELISA kits. Importantly, all laboratory personnel will be blinded to patients' characteristics and clinical outcomes, to ensure data quality and avoid observer bias.

Follow-ups and outcome determination

As the primary aim of this study is to determine the role of nasopharyngeal colonization in the development of CAP or IPD; after identifying patients colonized by S. pneumoniae during baseline experiments, patients will be followed every month by phone and every 6 months in our outpatient clinics to identify patients that develop CAP or IPD.

Patients will be asked to report any hospital visit (ER visit, hospital admission, and ICU admission) to the study coordinator and to bring discharge summaries provided by hospitals. Patients will be a follow-up for 2 consecutive years. During follow-ups, sample collection will be performed to determine whether patients develop nasopharyngeal colonization or change its systemic inflammatory profile. Samples will be collected and analyzed as baseline procedures.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age or older.
* Patients attending cardiology, pulmonology, endocrinology or rheumatology programs at the centers participating in the study.
* Patients with vaccination information available and confirmed in the medical records (in addition it will be confirmed at the time of the interview during the study enrollment consultation).
* Patients who sign the informed consent approved for this purpose.

Exclusion Criteria:

* Patients with a diagnosis of CAP prior to 90 days from the time of enrollment in the study.
* Patients admitted to hospital during the 7 days prior to enrollment in the study.
* Patients with any clinical or manifest limitation to provide biological samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients admitted to the outpatient service of 2 clinics in the city of Bogota D. C and at the Clínica Universitaria de la Sabana, who have been diagnosed with chronic diseases such as Heart Failure (HF), Benign Prostatic Hyperplasia (BPH), Chronic Cardiac Arrhythmia (CCA), Rheumatic Disease (RHD), bronchiectasis not related to cystic fibrosis, chronic obstructive pulmonary disease (COPD), among others; patients without evidence of pneumonia at study entry and who voluntarily approve their participation in the study will be recruited
Sampling Method: Probability Sample
Enrollment: 810 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Nasopharyngeal colonization by streptococcus pneumoniae | 2 years
  Definition: Colonization by S. pneumoniae in the nasopharyngeal tissue will be determined when using the traditional culture method and molecular biology (real time - PCR), the pneumococcus growth with a density of more than 10 (3) Colony-forming units (CFU).
  Then, using molecular biology (MS-PCR) and reaction quellung, S. pneumoniae isolated will be further characterized to determine the pneumococcal serotypes.
  Outcome measure:
  • Pneumococcal nasopharyngeal colonization prevalence of period in Adults With Chronic Diseases (PNCP) :
  PNCP = Pneumococcal isolates with bacteriological positive testing done during the study period / Total number of subjects enrolled in the study period.
  Statistic analysis: categorical variables will be expressed as counts (percentages), will be compared between groups using the Chi-squared test.

SECONDARY OUTCOMES:
Risk of Development of community-acquired pneumonia (CAP) | 2 years
  Definition: The analysis of the risk of developing CAP in adult subjects who are colonized in the nasopharynx with chronic diseases.
  Method: Patients will be followed-up by phone monthly and in-person every 6 months to determine whether they presented CAP or not.
  Outcome measure: Odds ratio (OR) of CAP in chronically ill adults who are colonized with pneumococcus in the nasopharynx (OR - NC).
  OR - CN = ((Cases of colonized subjects developing CAP) * (Non-colonized subjects that do not develop CAP))/((Colonized subjects that do not develop CAP) * (CAP cases of non-colonized patients with pneumococcal disease))
  Statistic analysis:
  * Regressions analyses.
  * Logistic regression.
  * A stratified analysis per comorbid condition (e.g., respiratory, cardiovascular, rheumatic, among others) will be carrying out.
  * Circular relation analysis.
  * A CHAID decision tree.
Risk of Development of Invasive Pneumococcal Disease (IPD) | 2 years
  Definition: IPD will be defined by the isolation of S pneumoniae from blood (bacteraemia) or cerebrospinal fluid (CSF; meningitis) in subjects by standard culture or PCR (Alanee et al., 2014; Aliberti et al., 2014; Reyes et al., 2017; Oldali et al., 2021).
  Outcome measure:
  Odds ratio (OR) of IPD in chronically ill adults who are colonized with pneumococcus in the nasopharynx (OR - IPD).
  OR - IPD = ((Cases of colonized subjects developing IPD) * (Non-colonized subjects that do not develop IPD))/((Colonized subjects that do not develop IPD) * (IPD cases of non-colonized patients with pneumococcal disease))
  Statistic analysis: Similar to the previous point, Regressions and Logistic regression analyses, A stratified analysis per comorbid condition will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Poveda, MD, Spc., Fellow, Study Chair — Fundación Clinica Abood Shaio
Locations (1):
- Clinica Universidad De La Sabana, Chía, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No
Confidentiality agreement